CLINICAL TRIAL: NCT00004416
Title: Randomized Study of Botulinum Toxin Type A for Achalasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: 199/13308; UTMB-FDR001421; JHH-94122903; MCMASTER-FDA; UTMB-97-230; UTMB-BB; UTMB-GCRC-470
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2001-04

CONDITIONS: Esophageal Achalasia
Keywords: achalasia; gastrointestinal disorders; rare disease
MeSH Terms: conditions — Esophageal Achalasia; Gastrointestinal Diseases; Rare Diseases | interventions — Botulinum Toxins, Type A

INTERVENTIONS:
Drug: botulinum toxin type A

SUMMARY:
OBJECTIVES: I. Compare the efficacy of two doses of botulinum toxin in the treatment of achalasia.

II. Compare the safety of these two doses in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, dose response study. Patients are randomized to one of two treatment arms; each arm receives a different dose of botulinum toxin type A.

All patients undergo a flexible upper gastrointestinal endoscopy. Botulinum toxin is injected into the lower esophageal sphincter into each of 4 quadrants. Some patients may receive a second treatment, depending on response and/or time of relapse.

Patients are followed daily for 7 days, then every 1-6 months for 1-2 years after treatment.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Diagnosis of achalasia by esophageal manometry and upper endoscopy
* Symptomatic including dysphagia, regurgitation, etc.
* No esophageal ulcers, Barrett's esophagus, significant esophagitis, or esophageal varices

--Patient Characteristics--

* Hematopoietic: Platelet count at least 50,000/mm3
* Hepatic: PT no greater than 3 seconds No severe hepatic problems
* Renal: No severe renal problems
* Cardiovascular: No recent myocardial infarction No unstable angina No decompensated congestive heart failure
* Pulmonary: No severe pulmonary disease with dyspnea at rest
* Other: No altered mental status No serious systemic disease Not pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56
Dates: Start 1997-01; Study Completion 2002-03

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Jay Pasricha, Study Chair — University of Texas